CLINICAL TRIAL: NCT01217606
Title: Safety and Efficacy of Triple Combination Therapy in Patients With Primary Open-Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 192024-062
Record Dates: First submitted 2010-10-07; First posted 2010-10-08 (Estimated); Results first posted 2015-11-09 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-11

CONDITIONS: Glaucoma, Open-Angle; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Bimatoprost; Brimonidine Tartrate, Timolol Maleate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Triple Combination Therapy (Experimental): Triple Combination Therapy with bimatoprost/brimonidine tartrate/timolol ophthalmic solution. One drop of Triple Combination Therapy administered to each eye, twice daily for up to 12 months.
  Interventions: Drug: bimatoprost/brimonidine tartrate/timolol ophthalmic solution (Triple Combination Therapy)
- Combigan® (Active Comparator): Fixed Combination brimonidine tartrate/timolol ophthalmic solution (Combigan®). One drop of Fixed Combination 0.2% brimonidine tartrate/0.5% timolol ophthalmic solution administered to each eye, twice daily for up to 12 months.
  Interventions: Drug: Fixed Combination 0.2% brimonidine tartrate/0.5% timolol ophthalmic solution

INTERVENTIONS:
Drug: bimatoprost/brimonidine tartrate/timolol ophthalmic solution (Triple Combination Therapy) — One drop of Triple Combination Therapy administered to each eye, twice daily for up to 12 months.
  Arms: Triple Combination Therapy
Drug: Fixed Combination 0.2% brimonidine tartrate/0.5% timolol ophthalmic solution — One drop of Fixed Combination 0.2% brimonidine tartrate/0.5% timolol ophthalmic solution administered to each eye, twice daily for up to 12 months.
  Other Names: COMBIGAN®
  Arms: Combigan®

SUMMARY:
This study will evaluate the safety and efficacy of Triple Combination Therapy compared with Fixed Combination brimonidine tartrate/timolol ophthalmic solution in patients with primary open-angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Ocular hypertension or primary open-angle glaucoma in each eye
* Requires treatment with IOP-lowering medication in both eyes

Exclusion Criteria:

* Required chronic use of ocular medications during the study other than study medication
* Use of any corticosteroids within 30 days
* History of any traumatic eye surgeries
* Cataract surgery in the past 6 months
* Anticipated wearing of contact lenses during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2011-01; Primary Completion 2014-09 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Belfort R Jr, Paula JS, Lopes Silva MJ, Della Paolera M, Kim T, Chen MY, Goodkin ML. Fixed-combination Bimatoprost/Brimonidine/Timolol in Glaucoma: A Randomized, Masked, Controlled, Phase III Study Conducted in Brazil☆. Clin Ther. 2020 Feb;42(2):263-275. doi: 10.1016/j.clinthera.2019.12.008. Epub 2020 Feb 20. PMID 32089329

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients were randomized into a 12-week Initial Treatment phase. Following this phase, patients may have continued into the 9-month Masked Extension on the same treatment assignment.
Groups:
- Triple Combination Therapy: Triple Combination Therapy with bimatoprost/brimonidine tartrate/timolol ophthalmic solution. One drop of Triple Combination Therapy administered to each eye, twice daily for 12 weeks in the Initial Treatment Phase followed by a 9 month Masked Extension.
- Combigan®: Fixed Combination brimonidine tartrate/timolol ophthalmic solution (Combigan®). One drop of Fixed Combination 0.2% brimonidine tartrate/0.5% timolol ophthalmic solution administered to each eye, twice daily for 12 weeks in the Initial Treatment Phase followed by a 9 month Masked Extension.
Period: Initial Treatment Phase
Arm/Group | Triple Combination Therapy | Combigan®
Started | 90 | 95
Completed | 76 | 83
Not Completed | 14 | 12
Not completed — Other Reasons | 0 | 2
Not completed — Protocol Violation | 3 | 2
Not completed — Personal Reasons | 0 | 2
Not completed — Lack of Efficacy | 1 | 0
Not completed — Adverse Event | 10 | 6
Period: 9-Month Masked Extension
Arm/Group | Triple Combination Therapy | Combigan®
Started | 67 | 73
Not Enrolled in Masked Extension | 9 | 10
Completed | 54 | 62
Not Completed | 13 | 11
Not completed — Adverse Event | 3 | 6
Not completed — Other Reasons | 4 | 4
Not completed — Personal Reasons | 2 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Pregnancy | 1 | 0
Not completed — Lack of Efficacy | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Triple Combination Therapy | Combigan® | Total
Number analyzed (Participants) | 90 | 95 | 185
Age, Customized [Number; unit: Participants]
  ≤65 years | 68 | 62 | 130
  >65 years | 22 | 33 | 55
Gender [Count of Participants; unit: Participants]
  Female | 53 | 63 | 116
  Male | 37 | 32 | 69

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Worse Eye Intraocular Pressure (IOP) Analyzed by Two-Sample T-Test
Description: Intraocular pressure (IOP) is a measurement of the fluid pressure inside the eye. IOP is evaluated at Hour 0 and Hour 2 in the worse eye, defined as the eye with the worse (higher) Hour 0 IOP at baseline. The mean of Hours 0 and 2 is calculated at Baseline and Week 12 in the worse eye. A negative number change from baseline indicates a reduction in IOP (improvement) and a positive number change from baseline indicates an increase in IOP (worsening). Data are analyzed using a two-sample t-test.
Time Frame: Baseline, Week 12
Population: Modified Intent to Treat: all randomized patients with at least one post-baseline efficacy evaluation
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury (mmHg)
Arm/Group | Triple Combination Therapy | Combigan®
Number analyzed (Participants) | 90 | 95
Millimeters of Mercury (mmHg)
  Baseline | 25.42 (2.902) | 24.43 (2.592)
  Change from Baseline at Week 12 (N=85, 93) | -10.45 (3.175) | -8.28 (3.256)

2. Secondary Outcome: Change From Baseline in Mean Worse Eye Intraocular Pressure (IOP) Analyzed by Mixed-Effect Model for Repeated Measure
Description: Intraocular pressure (IOP) is a measurement of the fluid pressure inside the eye. IOP is evaluated at Hour 0 and Hour 2 in the worse eye, defined as the eye with the worse (higher) Hour 0 IOP at baseline. The mean of Hours 0 and 2 is calculated at Baseline and Week 12 in the worse eye. A negative number change from baseline indicates a reduction in IOP (improvement) and a positive number change from baseline indicates an increase in IOP (worsening). Data are analyzed by a mixed-effect model for repeated measure.
Time Frame: Baseline, Week 1, Week 2, Week 4, Week 8, Week 12, Month 6, Month 9, Month 12
Population: Modified Intent to Treat: all randomized patients with at least one post-baseline efficacy evaluation and who have data at the noted time point (no missing imputation)
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury (mmHg)
Arm/Group | Triple Combination Therapy | Combigan®
Number analyzed (Participants) | 90 | 95
Millimeters of Mercury (mmHg)
  Baseline | 25.42 (2.902) | 24.43 (2.592)
  Change from Baseline at Week 1 (N=82, 91) | -11.63 (3.060) | -8.13 (2.969)
  Change from Baseline at Week 2 (N=82, 87) | -11.24 (3.283) | -8.12 (2.942)
  Change from Baseline at Week 4 (N=82, 88) | -10.88 (3.193) | -8.35 (3.100)
  Change from Baseline at Week 8 (N=75, 87) | -10.53 (3.165) | -7.94 (3.453)
  Change from Baseline at Week 12 (N=76, 83) | -10.56 (3.224) | -8.16 (3.161)
  Change from Baseline at Month 6 (N=64, 69) | -10.41 (2.976) | -8.29 (3.221)
  Change from Baseline at Month 9 (N=58, 67) | -10.29 (3.275) | -8.14 (2.937)
  Change from Baseline at Month 12 (N=55, 63) | -9.38 (3.398) | -7.58 (3.486)

3. Secondary Outcome: Change From Baseline in Mean Worse Eye Intraocular Pressure (IOP) Analyzed by Analysis of Covariance (ANCOVA)
Description: Intraocular pressure (IOP) is a measurement of the fluid pressure inside the eye. IOP is evaluated at Hour 0 and Hour 2 in the worse eye, defined as the eye with the worse (higher) IOP at baseline. The mean of Hours 0 and 2 is calculated at Baseline and Week 12 in the worse eye. A negative number change from baseline indicates a reduction in IOP (improvement) and a positive number change from baseline indicates an increase in IOP (worsening). Data are analyzed by ANCOVA.
Time Frame: Baseline, Week 1, Week 2, Week 4, Week 8, Week 12, Month 6, Month 9, Month 12
Population: Modified Intent to Treat: all randomized patients with at least one post-baseline efficacy evaluation
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury (mmHg)
Arm/Group | Triple Combination Therapy | Combigan®
Number analyzed (Participants) | 90 | 95
Millimeters of Mercury (mmHg)
  Baseline | 25.42 (2.902) | 24.43 (2.592)
  Change from Baseline at Week 1 (N=82, 91) | -11.63 (3.060) | -8.13 (2.969)
  Change from Baseline at Week 2 (N=84, 92) | -11.20 (3.290) | -8.28 (3.076)
  Change from Baseline at Week 4 (N=85, 93) | -10.85 (3.180) | -8.53 (3.228)
  Change from Baseline at Week 8 (N=85, 93) | -10.44 (3.105) | -8.07 (3.521)
  Change from Baseline at Week 12 (N=85, 93) | -10.45 (3.175) | -8.28 (3.256)
  Change from Baseline at Month 6 (N=67, 73) | -10.32 (2.965) | -8.42 (3.252)
  Change from Baseline at Month 9 (N=67, 73) | -10.09 (3.349) | -8.17 (3.031)
  Change from Baseline at Month 12 (N=67, 73) | -9.36 (3.368) | -7.77 (3.489)

ADVERSE EVENTS:
Description: Advers events (AEs) and serious adverse events (SAEs) are reported for the Safety Population. The Safety Population included all treated patients who received at least 1 dose of the study medication and attended at least 1 post-baseline visit.
Arm/Group | Triple Combination Therapy | Combigan®
Serious Adverse Events (participants affected / at risk) | 1/90 | 1/95
Other Adverse Events (participants affected / at risk) | 84/90 | 77/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Triple Combination Therapy (N=90) | Combigan® (N=95)
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Triple Combination Therapy (N=90) | Combigan® (N=95)
Conjunctival hyperaemia (Eye disorders) | 54 | 28
Punctate keratitis (Eye disorders) | 25 | 19
Eye pruritus (Eye disorders) | 12 | 7
Blepharitis (Eye disorders) | 15 | 12
Erythema of eyelid (Eye disorders) | 9 | 7
Eye irritation (Eye disorders) | 11 | 3
Conjunctival follicles (Eye disorders) | 7 | 15
Meibomianitis (Eye disorders) | 10 | 8
Eye allergy (Eye disorders) | 6 | 5
Cataract (Eye disorders) | 8 | 3
Visual Field Defect (Nervous system disorders) | 7 | 7
Blepharal Pigmentation (Eye disorders) | 6 | 1
Hypertrichosis (Skin and subcutaneous tissue disorders) | 5 | 2
Influenza (Infections and infestations) | 5 | 2
Visual Acuity Reduced (Eye disorders) | 5 | 1
Pinguecula (Eye disorders) | 4 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.